CLINICAL TRIAL: NCT07215663
Title: A Phase 1b, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Systemic Lupus Erythematosus
Brief Title: Clinical Study of Cizutamig in Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Candid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND106-103
Record Dates: First submitted 2025-09-23; First posted 2025-10-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cizutamig (Experimental)
  Interventions: Drug: Cizutamig

INTERVENTIONS:
Drug: Cizutamig — Cizutamig will be dosed according to the protocol
  Other Names: CND106

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK, PD, immunogenicity, and preliminary clinical activity of Cizutamig in patients with Systemic Lupus Erythematosus

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary clinical activity of cizutamig in patients with Systemic Lupus Erythematosus

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old at the time of signing the informed consent form
2. Diagnosis of SLE according to the ACR/EULAR classification criteria
3. Positive anti-dsDNA or positive anti-Smith antibodies AND positive for at least one other of anti-dsDNA, anti-Smith antibodies, or ANA ≥1:80 at screening
4. SLEDAI-2K total score ≥6 and SLEDAI-2K clinical score≥4 at Screening
5. The investigator judged that the patient had an inadequate response to prior treatment for at least 3 months before screening
6. Stable use of concomitant therapies
7. For patients with active LN only: LN Class III or IV

Exclusion Criteria:

1. Inadequate clinical laboratory parameters at Screening
2. Active infection
3. Receipt of or inability to discontinue any excluded therapies
4. Receipt of live vaccine within 4 weeks prior to Screening
5. Presence of any concomitant autoimmune disease
6. Active or known history of catastrophic anti-phospholipid syndrome (APS)
7. APS or thrombotic event not adequately controlled by anticoagulation therapy
8. History of progressive multifocal leukoencephalopathy
9. History of primary immunodeficiency or a hereditary deficiency of the complement system
10. Central nervous system disease
11. Presence of 1 or more significant concurrent medical conditions
12. Have a diagnosis or history of malignant disease within 5 years
13. Serious mental illness, alcohol or drug abuse, dementia, or any other condition that would impair the patient's ability to receive the planned treatment or to understand informed consent at the study site as determined by local practice
14. Inability to comply with protocol-mandated requirements
15. History of severe allergic or anaphylactic reactions to mAb therapy (or recombinant antibody-related fusion proteins) or any constituents of cizutamig
16. History of or planned organ transplant and/or autologous or allogeneic hematopoietic stem cell transplantation
17. Major surgery requiring use of general anesthesia within 12 weeks or planned or expected major surgery during the study
18. Women who are pregnant or breastfeeding
19. Patients who do not agree to the use of highly effective contraception as defined by the protocol
20. Individuals considered to be part of a vulnerable population (eg, incarceration)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events through end of study | Baseline to Month 12
Changes from baseline in vital signs through end of study: body temperature | Baseline to Month 12
Changes from baseline in vital signs through end of study: heart rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: respiratory rate | Baseline to Month 12
Changes from baseline in vital signs through end of study: blood pressure | Baseline to Month 12
Changes from baseline in vital signs through end of study: pulse oximetry | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: PR interval | Baseline to Month12
Changes from baseline in ECG parameters through end of study: QRS interval | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: QTcF interval | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: serum chemistry | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study: hematology | Baseline to Month 12

SECONDARY OUTCOMES:
Pharmacokinetic (PK) for Cizutamig: Cmax | Baseline to Month 12
PK parameters for Cizutamig: time of maximum concentration | Baseline to Month 12
PK parameters for Cizutamig: area under the concentration-time curve | Baseline to Month 12
PK parameters for Cizutamig: clearance | Baseline to Month 12
PK parameters for Cizutamig: volume of distribution | Baseline to Month 12
PK parameters for Cizutamig: half-life | Baseline to Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No